CLINICAL TRIAL: NCT05037032
Title: Effects of Naltrexone on Nocturnal Breathing Patterns at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, James D. Anholm, M.D., Staff physician; Pulmonary & Critical Care, VA Loma Linda Health Care System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1392
Record Dates: First submitted 2021-08-20; First posted 2021-09-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Altitude; Sleep Apnea, Central
Keywords: Altitude; Periodic Breathing; Sleep
MeSH Terms: conditions — Sleep Apnea, Central | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized double-blind, placebo controlled crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug naltrexone hydrochloride (Active Comparator): 50 mg Naltrexone PO
  Interventions: Drug: Naltrexone Pill
- Matching placebo for naltrexone hydrochloride (Placebo Comparator): Matching placebo for Study Drug Naltrexone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone Pill — 50 mg PO one-time only
  Arms: Study drug naltrexone hydrochloride
Drug: Placebo — Matching placebo for naltrexone
  Arms: Matching placebo for naltrexone hydrochloride

SUMMARY:
Sleep at altitude is often poor. The purpose of this study is to evaluate the effects of a single dose of the opioid antagonist, naltrexone, on sleep quality and periodic breathing after rapid ascent to ~3800m altitude.

DETAILED DESCRIPTION:
Sleep at high altitude is notoriously poor due to a combination of the unusual sleep environment and hypoxia during sleep. Many people develop what is called periodic breathing (PB) during sleep. PB may improve overall mean nocturnal oxygen saturation (SpO2) although this is not entirely clear. Simultaneously, PB may further disturb sleep at altitude and has been associated with nighttime arousals from sleep. Medications that may decrease the amount of PB might improve sleep quality. The FDA approved drug, naltrexone, is a specific antagonist to the brain opioid receptors. It is a non-addicting drug which has never been studied at altitude.

Clinical Relationships: Sleep disordered breathing is a very common disorder throughout the population, but it worsens with increasing age and BMI. At the same time, many in our Veteran population live in the local mountains and undoubtedly develop PB during sleep in addition to having obstructive sleep apnea.

Objectives: The purpose to this study is to evaluate the effects of a single dose of naltrexone on PB and oxygen saturation during sleep at altitude in healthy young participants. The additional purpose will be to assess the subject-perceived sleep quality after the use of naltrexone vs. placebo.

Research Design: A prospective, randomized, double-blind, crossover study.

Methodology: We plan recruit up to 30 healthy study subjects with no history of sleep disordered breathing. Potential participants will be screened to ensure inclusion and exclusion criteria are met. A baseline low altitude sleep study will be preformed at home. No medication will be given before this baseline sleep study. The sleep study will be similar to the home sleep studies routinely used by the VA Loma Linda Healthcare System's Sleep Center. Participants will be transported for High Altitude Trip 1 to the Barcroft Laboratory at the White Mountain Research Center (WMRC) at 3810 m altitude. At WMRC they will have a sleep study performed, similar to the baseline sleep study, after taking either a single dose of naltrexone or matching placebo. After an appropriate washout period (at least 5 half-lives) subjects will again be studied (High Altitude Trip 2) taking the alternate medication (naltrexone/placebo) to the one used in the first study. Order of placebo vs. naltrexone will be randomized. Prior to sleep the subject will fill out questionnaires detailing how sleepy they are. On the morning following each sleep study, subjects will fill out a short questionnaire assessing the quality of their sleep.

Impact/Significance: Improved knowledge of the mechanisms of PB in hypoxic environments will provide important insights into diagnostic and therapeutic decisions for Veterans who suffer from sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females
2. Age 18 to 35 years of age
3. Body-mass index (BMI) ≤ 27
4. At least two weeks after full vaccination for Sars-CoV-2. Proof of vaccination will be determined by the investigators.

Exclusion Criteria:

1. Current smoker or significant past smoking history (≥ 10 pack-years)
2. History of COPD, interstitial lung disease or other pulmonary disease that in the opinion of the investigators would compromise the subject's safety at altitude
3. History of obstructive sleep apnea, or other history of sleep disordered breathing, or previous use of nighttime continuous positive airway pressure (CPAP)
4. Any history of chronic opioid use or prior abuse history
5. Any history of alcohol abuse
6. Use of any opioid substance (prescribed or otherwise) within 2-weeks of study enrollment
7. Any medications that might, in the opinion of the investigators, interfere with or alter respiratory control, (e.g. acetazolamide). Use of oral contraceptive medications would be allowed as long as the study subject is on the same agent/dose during both arms of the study.
8. Recent (within 3 weeks) exposure to altitudes ≥ 3,500 m at time of 1st altitude trip

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Nighttime oxygen saturation | Up to 60 days
  Change from baseline in nighttime SpO2
Periodic Breathing | Up to 60 days
  Change from baseline in portion of night spent with periodic breathing
Epworth Sleepiness Scale | Up to 60 days
  Subjective measurement of one's daytime sleepiness (0 = less sleepy, 24= excessively sleepy)
Stanford Sleepiness Scale | Up to 60 days
  Self-reported assessments of how alert one is currently feeling (1= wide awake, X=asleep)
Groningen Sleep Quality Scale | Up to 60 days
  Assessment to understand sleep quality (0 = good sleep, maximum score of 14 points indicates poor sleep the night before)

CONTACTS AND LOCATIONS:
Overall Officials: James D Anholm, MD, Principal Investigator — VA Loma Linda Healthcare System
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No